CLINICAL TRIAL: NCT02766634
Title: A Randomized Open-label, Multiple-dose, Crossover Study Evaluatig The Pharmacodynamics And Pharmacokinetics Of Filgrastim Hospira Compared To Us-approved Neupogen (Registered) Following Subcutaneous Administration To Healthy Volunteers
Brief Title: A Research Study To Test How Multiple Doses Of Filgrastim Hospira Works In The Body Of Healthy Study Subjects When Given by Subcutaneous Injection (SC) (Shot) Compared To An Already U.S.-Approved Drug Neupogen® (Amgen)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ZIN-FIL-1501; C1121003 (Other: Alias Study Number)
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Neutropenia (Low White Blood Cell Count)
Keywords: filgrastim
MeSH Terms: conditions — Neutropenia; Leukopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Filgrastim Hospira (US) followed by U.S.-approved Neupogen® (Experimental)
  Interventions: Biological: Filgrastim Hospira (US); Biological: U.S.-approved Neupogen®
- U.S.-approved Neupogen® followed by Filgrastim Hospira (US) (Experimental)
  Interventions: Biological: Filgrastim Hospira (US); Biological: U.S.-approved Neupogen®

INTERVENTIONS:
Biological: Filgrastim Hospira (US) — 5 micrograms/kilogram (ug/kg) subcutaneous (SC) injection once a day for 5 days
Biological: U.S.-approved Neupogen® — 5 micrograms/kilogram (ug/kg) subcutaneous (SC) injection once a day for 5 days

SUMMARY:
This is a study comparing two study drugs, Filgrastim Hospira and Neupogen®. Neupogen® is approved by the US Food and Drug Administration (FDA) to treat low numbers of specific kinds of white blood cells (WBC) known as neutrophils. This type of white cell is important in fighting infections. A low neutrophil count is known as neutropenia. Both drugs work by increasing the number of neutrophils that are produced in the body.

This is important for patients who have low neutrophils due to chemotherapy, other treatments such as bone marrow transplant or certain other conditions with symptoms/problems related to low neutrophil counts. The main aim of the study is to test how Filgrastim Hospira works in the body compared to Neupogen®.

DETAILED DESCRIPTION:
This is a randomized, open-label, multiple-dose, crossover study evaluating the pharmacodynamics and Pharmacokinetics equivalence following SC administration of test and reference product in healthy volunteers. The study will be conducted at a single Phase 1 unit. There will be 30 healthy subjects in each of the two sequences.

After meeting the selection criteria, subjects will be randomly assigned to 1 of the 2 treatment sequences:

* Filgrastim Hospira (US) in Period 1 followed by US-approved Neupogen® in Period 2.
* US-approved Neupogen® in Period 1 followed by Filgrastim Hospira (US) in Period 2.

Subjects will receive one of each of the drugs once a day for 5 days in each of the treatment sequences.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for study participation if all of the following criteria are met at Screening:

1. Provides written informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB) prior to any study related activities
2. Healthy male or female volunteers between 18 and 65 years of age (both inclusive)
3. Body mass index (BMI) between 19 and 30 kg/m2, inclusive, and body weight of not < 50 kg or > 100 kg
4. Non smoker (defined as a subject who has not smoked and has not used nicotine containing products for at least 3 months prior to study drug administration and has a negative urine screen for cotinine) at Screening
5. Female subjects of childbearing potential and male subjects and their partners of childbearing potential, agree to pregnancy prevention throughout the duration of the study (through the Final Visit). Subjects and their partners must agree to use of an effective method of contraception, to avoid impregnation of females throughout the course of the study. Subjects using oral contraceptives must be on a stable regimen for at least 3 months prior to Screening. While the best way to avoid pregnancy is to abstain from sexual activity, adequate forms of contraception to be used include oral contraception, depot contraception, intrauterine device (IUD), and barrier contraceptive methods, such as condoms and barrier creams/contraceptive jellies, and spermicidals. Subjects and their partners who can become pregnant must use contraception while on study drug from admission to the Final Visit. Male subjects must also refrain from donating sperm from admission to the Final Visit
6. Agrees to abstain from alcohol consumption throughout duration of the study and has a negative urine for alcohol at Screening

Exclusion Criteria:

A subject will NOT be eligible for study participation if any of the following criteria are met at Screening:

1. Any active systemic or immunologic disease or condition, including but not limited to the following general categories: cardiovascular/pulmonary, hepatorenal, or systemic infection, or lactation
2. Hematologic laboratory abnormalities including leukocytosis (defined as total leukocytes > 11,000/µL), leukopenia (defined as total leukocytes < 4000/μL), or neutropenia (defined as absolute neutrophil count [ANC] < 1500/µL) or thrombocytopenia (defined as platelet count of < 150/µL)
3. Clinically significant, as judged by the Investigator, vital sign, chest X-ray, or 12-lead electrocardiogram (ECG) abnormality
4. History of biological growth factor exposure, including but not limited to filgrastim and other granulocyte-colony stimulating factors (G-CSFs) in the context of treatment, prophylaxis, peripheral blood stem cell mobilization, or previous investigational study setting
5. Drug sensitivity, allergic reaction to, or known hypersensitivity/idiosyncratic reaction to Escherichia coli-derived proteins, filgrastim, pegfilgrastim, other granulocyte colony-stimulating factors or any component of the product: Subjects with the rare heredity problem of fructose intolerance are excluded due to the excipient sorbitol
6. History of splenic rupture (or subject who is asplenic), pulmonary infiltrate or pneumonia, sickle cell disorders, chronic neutropenia, thrombocytopenia, or vasculitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The Area under the effect curve for CD34+ (AUECCD34+) | prior to study drug administration on Days 1, 2, 3, 4, 5, and 24, 48, 72, 96, and 120 hours after dose administration on Day 5 of each period
Maximum observed value for CD34+ (CD34+max) | prior to study drug administration on Days 1, 2, 3, 4, 5, and 24, 48, 72, 96, and 120 hours after dose administration on Day 5 of each period
Area under the serum filgrastim concentration versus time curve from time zero to 24 hours (AUC0-24) | prior to study drug administration and 24, 48, 72, 96, and 120 hours after dose administration on Day 5 of each period
Maximum serum filgrastim concentration (Cmax) following study drug administration on Day 5 | prior to study drug administration and 24, 48, 72, 96, and 120 hours after dose administration on Day 5 of each period

SECONDARY OUTCOMES:
Time to maximum CD34+ count (Tmax[CD34+]) | prior to study drug administration on Days 1, 2, 3, 4, 5, and 24, 48, 72, 96, and 120 hours after dose administration on Day 5 of each period
The concentration prior to dose on Day 5 (Ctrough) | prior to study drug administration and 24, 48, 72, 96, and 120 hours after dose administration on Day 5 of each period.
Time to maximum serum filgrastim concentration (Tmax) | prior to study drug administration and 24, 48, 72, 96, and 120 hours after dose administration on Day 5 of each period.
Elimination half-life (t1/2) from serum filgrastim concentrations following dose administration on Day 5 | prior to study drug administration and 24, 48, 72, 96, and 120 hours after dose administration on Day 5 of each period.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- SeaView Research, Inc., Miami, Florida, United States

REFERENCES:
- [Derived] Yao HM, Ottery FD, Borema T, Harris S, Levy J, May TB, Moosavi S, Zhang J, Summers M. PF-06881893 (Nivestym), a Filgrastim Biosimilar, Versus US-Licensed Filgrastim Reference Product (US-Neupogen(R)): Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Safety of Single or Multiple Subcutaneous Doses in Healthy Volunteers. BioDrugs. 2019 Apr;33(2):207-220. doi: 10.1007/s40259-019-00343-8. PMID 30900158
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=ZIN-FIL-1501&StudyName=A+Randomized+Open-label%2C+Multiple-dose%2C+Crossover+Study+Evaluatig+The+Pharmacodynamics+And+Pharmacokinetics+Of+Filgrastim+Hospira+Compared+To+Us-approved+Neupogen+%28registered%29+Following+Subcutaneous+Administration+To+Healthy+Volunteers